CLINICAL TRIAL: NCT02722031
Title: Severe Hypoxemia : Prevalence, Treatment and Outcome
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: SPECTRUM
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Critically Ill Patients Admitted in ICU
Keywords: intensive care; prevalence; hypoxemia; ARDS
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Hypoxemia is usually observed during ICU stay. Nevertheless, the prevalence of hypoxemia among patients admitted in ICU is not well known, in partly due to a lack of a consensual definition. Some of these patients meet the criteria of Acute Respiratory Distress Syndrome whom the definition has been recently modified in 2011. Many uncertainties are remaining in considering the patients with ARDS: prevalence of the category of "mild ARDS", the proportion of patients with invasive mechanical ventilation, the therapeutic modalities and the prognosis, in particular, the move towards a more severe ARDS category. Finally, many patients with hypoxemia do not meet ARDS definition. The prevalence of this population in ICU is unknown, likewise its prognosis. In this way, it would be interesting to compare, for each levels of hypoxemia (mild, moderate and severe) the prognosis of the patients with and without ARDS.

The main objective of the SPECTRUM study is to assess the prevalence of hypoxemia in French-speaking Intensive Care Unit in 2016 in using a single-day point-prevalence study design. Two periods of inclusion have been, actually, planned: from the 29th Mars to the 31st Mars and from the 5th to the 7th April. In each participating center, the day of the study will be chosen among these periods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Hospitalized in ICU during the 24 hours of the study
* Information provided to the patient or proxy

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Patient under guardianship or curators
* Lack of social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted in Intensive Care
Sampling Method: Non-Probability Sample
Enrollment: 1694 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypoxemia defined by a ratio of the Partial Pressure of Oxygen in Arterial Blood (PaO2) / Fraction of inspired oxygen (FiO2) below 300 mm Hg | 1 day
  prevalence of hypoxemia among patients hospitalized in ICU the day of the study

SECONDARY OUTCOMES:
Prevalence of severe hypoxemia defined by a ratio PaO2/ FiO2 below 100 mm Hg | 1 day
Prevalence of mild hypoxemia defined by a ratio PaO2/FiO2 below 200 mm Hg and above 100 mm Hg | 1 day
Prevalence of moderate hypoxemia defined by a ratio PaO2/FiO2 below 300 mm Hg and above 200 mm Hg | 1 day
Prevalence of Acute Respiratory Distress Syndrome (ARDS) according the Berlin definition | 1 day
ICU mortality | 90 days
Prevalence of the different modalities of oxygen therapy | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Bretonneau, Tours, France

REFERENCES:
- [Result] Linko R, Okkonen M, Pettila V, Perttila J, Parviainen I, Ruokonen E, Tenhunen J, Ala-Kokko T, Varpula T; FINNALI-study group. Acute respiratory failure in intensive care units. FINNALI: a prospective cohort study. Intensive Care Med. 2009 Aug;35(8):1352-61. doi: 10.1007/s00134-009-1519-z. Epub 2009 Jun 13. PMID 19526218
- [Result] Brun-Buisson C, Minelli C, Bertolini G, Brazzi L, Pimentel J, Lewandowski K, Bion J, Romand JA, Villar J, Thorsteinsson A, Damas P, Armaganidis A, Lemaire F; ALIVE Study Group. Epidemiology and outcome of acute lung injury in European intensive care units. Results from the ALIVE study. Intensive Care Med. 2004 Jan;30(1):51-61. doi: 10.1007/s00134-003-2022-6. Epub 2003 Oct 16. PMID 14569423
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Derived] SRLF Trial Group. Hypoxemia in the ICU: prevalence, treatment, and outcome. Ann Intensive Care. 2018 Aug 13;8(1):82. doi: 10.1186/s13613-018-0424-4. PMID 30105416